CLINICAL TRIAL: NCT03624543
Title: A Phase II Study of CFI-400945 in Patients With Advanced/Metastatic Breast Cancer
Brief Title: CFI-400945 in Patients With Advanced/Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Stand Up To Cancer Canada-Canadian Cancer Society Breast Cancer Dream Team (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I237
Record Dates: First submitted 2018-08-01; First posted 2018-08-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 2-(3-(4-((2,6-dimethylmorpholino)methyl)styryl)-1H-indazol-6-yl)-5'-methoxyspiro(cyclopropane-1,3'-indolin)-2'-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: TNBC (Experimental): N=9 to 24 patients
  Interventions: Drug: CFI-400945
- Cohort 2: PTEN-null, ER+ and/or PR+, HER2- (Experimental): N=9 to 24 patients
  Interventions: Drug: CFI-400945
- Cohort 3: Not PTEN-null, ER+ and/or PR+, HER2- (Experimental): N=9 to 24 patients
  Interventions: Drug: CFI-400945

INTERVENTIONS:
Drug: CFI-400945 — 32mg; 28 day cycles; Cycle 1: Days 1-7 then 15-21 Cycle 2 onward: Daily

SUMMARY:
The standard or usual treatment for this disease is to undergo chemotherapy to slow the spread of the disease and relieve some symptoms of cancer. Patients will have already had at least one chemotherapy treatment for their disease at this stage.

DETAILED DESCRIPTION:
CFI-400945 is a new type of drug for breast cancer. Laboratory tests show that it works by blocking a specific protein called Polo-like Kinase 4 (PLK4) that is involved in cancer cell growth. CFI-400945 may slow down the growth of cancer cells or may cause cancer cells to die. This drug has been shown to shrink tumours in animals and has been studied in some patients and appears well tolerated with little side effects. CFI-400945 seems promising but it is not clear if it can offer better results than standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically and/or cytologically confirmed diagnosis of breast cancer, that is advanced/metastatic/recurrent or unresectable, for which no curative therapy exists, either:

  * Negative for ER, PR and HER2 by ASCO/CAP criteria (COHORT 1) OR
  * Positive for ER and or PR and negative for HER2 AND

    * loss or mutation of PTEN, as assessed by IHC assay (COHORT 2) OR
    * No loss or mutation of PTEN, as assessed by IHC assay (COHORT 3)

For the patients entered on the PK/safety component only, results of the PTEN status may be documented after enrollment

* Only female patients will be enrolled.
* All patients must have a formalin fixed paraffin embedded tissue block (from primary or metastatic tumour) available and must have provided informed consent for the release of the block. Biopsies are optional but strongly encouraged for patients with accessible disease suitable for biopsy. The timing of tumour biopsies for patients who provide informed consent and willing is prior to treatment (after enrollment), and again between cycle 2 day 15- day 22. An additional biopsy at the time of progression in patients with clinical benefit is also encouraged. Lesions planned for biopsy may not be the only target lesion.
* Presence of clinically and/or radiologically documented disease. All radiology studies must be performed within 21 days prior to enrollment (within 28 days if negative).
* All patients must have measurable disease as defined by RECIST 1.1. The criteria for defining measurable disease are as follows: Chest x-ray ≥ 20 mm CT scan (with slice thickness of 5 mm) ≥ 10 mm --> longest diameter Physical exam (using calipers) ≥ 10 mm Lymph nodes by CT scan ≥ 15 mm --> measured in short axis
* Patients must be ≥ 18 years of age.
* Patients must have an ECOG performance status of 0 or 1.
* Patients must have a life expectancy of 3 months or longer.
* Laboratory Requirements (must be done within 7 days prior to enrollment) Absolute neutrophils ≥ 1.5 x 10^9/L Platelets ≥ 100 x 10^9/L Bilirubin ≤ 1.5 x ULN (upper limit of normal) AST and ALT ≤ 2.5 x ULN; ≤ 4.0 x ULN if patient has liver metastases Serum creatinine ≤ 1.5 x ULN or Creatinine clearance ≥ 50 mL/min
* Patients must be able to swallow oral medications and have no known gastrointestinal disorders that may interfere with absorption (such as malabsorption).
* Patients must have had at least 1 prior line of cytotoxic chemotherapy for breast cancer, in any setting, which must have included an anthracycline and a taxane (unless contraindicated). Select patients that have not received both anthracycline and taxane therapy may be considered eligible after discussion with CCTG. There is no limit to the number of prior chemotherapy regimens
* Patients may have received other therapies including endocrine therapy, immunotherapy, and/or targeted therapies (including CDK4/6 inhibitors).
* Patients must have recovered (to at least grade 0 or 1) from all reversible toxicity related to prior chemotherapy or systemic therapy and have adequate washout as follows:
* Longest of one of the following:

  * Two weeks,
  * 5 half-lives for investigational agents
  * Standard cycle length of standard therapies.
* Prior external beam radiation is permitted provided a minimum of 28 days (4 weeks) have elapsed between the last dose of radiation and date of enrollment. Exceptions may be made for low-dose, non-myelosuppressive radiotherapy after consultation with CCTG. Concurrent radiotherapy is not permitted.
* Previous surgery is permitted provided that a minimum of 21 days (3 weeks) have elapsed between any major surgery and date of enrollment and that wound healing has occurred.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Patients must be accessible for treatment and follow up. Patients enrolled on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial.
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of patient enrollment.
* Women of childbearing potential must have agreed to use a highly effective contraceptive method

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for > 2 years and which do not require ongoing treatment.
* Patients with active or uncontrolled infections or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol.
* Patients are not eligible if they have a known hypersensitivity to the study drug(s) or their components.
* Patients with HER2 positive breast cancer (based on the most recent assessment).
* Patients with significant cardiac (including uncontrolled hypertension) or pulmonary disease, or active CNS disease or infection. Patients should have a LVEF ≥ 50%.
* Patients may not receive concurrent treatment with other anti-cancer therapy (other than bone-targeted therapy, if already taking and stable) or investigational agents while on protocol therapy.
* Patients who have received growth factors within 28 days prior to initiation of dosing of CFI-400945 or who will require treatment with growth factors throughout the duration of the trial.
* Pregnant or breastfeeding women.
* Patients being treated with drugs listed in Appendix V Table 1 are excluded. Patients being treated with drugs listed in Appendix V Table 2 may be enrolled, but should be monitored carefully for toxicities resulting from potential interactions between CFI-400945m and these drugs. In addition, patients must avoid consumption of the fruit or juice of Seville oranges (e.g. marmalade), grapefruit, pomelos and star fruit from 7 days before the first dose of study drug and during the entire study due to potential CYP3A4 interaction with the study drug. Regular orange juice is allowed.
* Patients with history of central nervous system metastases or spinal cord compression unless they have received definitive treatment, are clinically stable and do not require corticosteroids.
* Patients with any medical condition that would impair the administration of oral agents including significant bowel resection, inflammatory bowel disease or uncontrolled nausea or vomiting.
* Patients being treated with full dose warfarin. Patients with history of deep vein thrombosis or pulmonary embolus who are being treated with therapeutic doses of low molecular weight heparin, direct factor Xa inhibitors or prophylactic dose anticoagulants may be enrolled

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 51 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response defined by RECIST 1.1 | 2 years

SECONDARY OUTCOMES:
Disease Control Rate (DCR) defined by RECIST 1.1 | 2 years
Number and severity of adverse events | 2 years
Molecular analyses of CFI-400945 on tumour cells through paired tumour biopsies using next generation DNA sequencing | 2 years
  Molecular analyses including next-generation DNA sequencing will be performed on archival and recent tumour (or normal tissue) materials to identify potential biomarkers of response, histologically assess centrosomes and aberrant mitoses, and evaluate genomic alterations and other molecular features (i.e. gene or protein expression levels).
Molecular analyses of CFI-400945 on tumour cells through paired biopsies using immunohistochemistry | 2 years
  Assessment of centrosomes and aberrant mitoses and evaluation of genomic alterations and other molecular features (i.e. gene or protein expression levels) by molecular analyses including immunohistochemistry performed on archival and recent tumour (or normal tissue) materials to identify potential biomarkers of response.

CONTACTS AND LOCATIONS:
Overall Officials: David Cescon, Study Chair — Princess Margaret Cancer Centre, Toronto, ON; Rossanna Pezo, Study Chair — Sunnybrook Health Sciences Centre, Toronto, ON
Locations (6):
- Canada (6):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No